CLINICAL TRIAL: NCT07186244
Title: Implementation of an Italian Cohort of People on HIV-1 Pre-exposure Prophylaxis Within the ICONA Network: PrIDE (Prevention ICONA Dedicated Ensemble)
Brief Title: Prevention ICONA Dedicated Ensemble
Acronym: PrIDE
Status: Recruiting | Type: Observational
Sponsor: Fondazione ICONA (Other)
Responsible Party: Sponsor
Other Study IDs: 1539
Record Dates: First submitted 2025-08-04; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: PrEP; PrEP Adherence Monitoring; HIV; HIV -1 Infection; STI; STI Prevention
Keywords: PrEP; HIV; STI; STI Prevention
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants who experience a documented HIV seroconversion (breakthrough infection) during the study or within 12 months after its completion, defined as reactivity to a 4th-generation HIV Ab/Ag test with detectable HIV-RNA on real-time PCR testing, will undergo blood sampling for:
  * Pharmacological drug level testing in peripheral blood
  * Lymphocyte typing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- PrIDE Cohort

SUMMARY:
Despite significant advances in HIV treatment, transmission remains a public health concern. In 2022, there were 1.3 million new HIV infections worldwide and 1,888 new diagnoses in Italy, with sexual transmission being the predominant route. Many individuals are still diagnosed late, and a portion of people living with HIV are unaware of their status. Pre-Exposure Prophylaxis (PrEP) has emerged as an effective biomedical strategy to prevent new infections, especially when integrated into comprehensive prevention efforts.

Study Objectives The primary objective of this observational study is to establish a large prospective cohort of individuals using PrEP in Italy. The study aims to assess PrEP's effectiveness, tolerability, adherence, and barriers to long-term use in a real-world setting. These data will be instrumental in guiding future strategic interventions to optimize PrEP management and move toward the goal of zero new HIV infections in Italy.

Primary Objective

* To assess the incidence of new HIV infections among PrEP users in Italy. Secondary Objectives
* Incidence of other sexually transmitted infections (STIs);
* Tolerability of PrEP;
* Psychological and behavioral aspects related to PrEP use;
* Adherence and persistence in care;
* Use of therapies and prophylaxis for STIs during PrEP use. Study Design and Coordination This is a prospective observational study, promoted by Fondazione ICONA in collaboration with clinical centers and community-based organizations. The coordinating enrolling center is INMI "L. Spallanzani" IRCCS in Rome.

Participating Centers:

* 49 university and hospital-based centers across Italy;
* 4 non-clinical checkpoints offering PrEP screening, prescription, and follow-up.

Study Population Adults (≥18 years) who are HIV-negative, sexually active, and considered eligible for PrEP per national or international guidelines, including both new and current PrEP users.

Inclusion Criteria

* Age ≥18 years;
* Negative HIV test at enrollment;
* Willingness to initiate or continue PrEP;
* Informed consent provided. Exclusion Criteria
* HIV infection or strong suspicion of infection;
* Contraindications to PrEP medications; Known allergy to PrEP components; Refusal to comply with study procedures.

DETAILED DESCRIPTION:
The PrIDE study is a national, multicenter, prospective observational cohort aimed at assessing the effectiveness and real-world implementation of HIV pre-exposure prophylaxis (PrEP) in Italy. It collects sociodemographic, clinical, laboratory, behavioral, and quality-of-life data from about 5,000 HIV-negative adults (≥18 years) initiating or already on PrEP, in accordance with Italian and international guidelines.

All 49 university and hospital infectious disease clinics and 4 community-based checkpoints across Italy can participate. Participants are followed every 3-5 months through routine clinical visits, including HIV/STI testing, safety labs, and electronic questionnaires via a dedicated mobile app.

The primary objective is to estimate the incidence of HIV seroconversion, while secondary aims include monitoring sexually transmitted infections, evaluating safety and tolerability, and analyzing adherence, persistence, and behavioral factors. Data are collected in a secure, encrypted eCRF managed by the ICONA Foundation.

The study is coordinated by the National Institute for Infectious Diseases "L. Spallanzani" IRCCS in Rome, will run for at least 10 years, and requires approval from the Ethics Committees of all participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Negative HIV Ab/Ag test (4th generation or higher) at the enrollment visit
* Request and/or willingness to take PrEP, or already on PrEP
* Ability to understand the study procedures and to sign informed consent

Exclusion Criteria:

* Individuals with HIV infection or with strong clinical/epidemiological suspicion of HIV infection
* Individuals with contraindications to the use of medications included in the PrEP regimen (as per the product information)
* Documented allergy to one or more pharmacological components of the proposed PrEP regimen
* Lack of willingness to adhere to the required procedures and follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective enrollment is planned for all individuals taking PrEP in Italy, with the aim of establishing a cohort under active follow-up.
  Eligible participants are adults (>18 years old), HIV-negative, and sexually active, who-according to approved national and international guidelines and/or standard clinical practice-are deemed suitable to receive a PrEP prescription or are already undergoing PrEP.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of HIV seroconversion in individuals taking PrEP, from the time of cohort enrollment. | Perioperative/Periprocedural
  HIV seroconversion is defined as a new HIV infection occurring in a participant during the observational follow-up period. Seroconversion will be determined by a reactive 4th-generation HIV antibody/antigen (Ab/Ag) test confirmed by detectable HIV-RNA using real-time PCR. The measure will be taken at routine clinical visits approximately every 3 months, or when clinically indicated, according to national guidelines. All cases of confirmed HIV infection will be reviewed and documented by the coordinating center.

SECONDARY OUTCOMES:
Tolerability of PrEP expressed as the number of adverse events per person-years of follow-up after study enrollment | Perioperative/Periprocedural
Assess behavioral-related factors influencing PrEP use and persistence in care through questionnaires | Perioperative/Periprocedural
  Values monitored through ePROs questionnaire completed by participants at each visit.
Assess adherence-related factors influencing PrEP use and persistence in care through questionnaire | Perioperative/Periprocedural

CONTACTS AND LOCATIONS:
Locations (53):
- Italy (53):
  - Ospedale Clinicizzato SS. Annunziata - Scuola di Specializzazione di Malattie Infettive, Chieti, Abruzzo
  - Ospedale Civile Santo Spirito - U.O. Malattie Infettive, Pescara, Abruzzo
  - AOU Consorziale - Policlinico Giovanni XXIII - Struttura Complessa di Malattie Infettive, Bari, Apulia
  - A.O.U. Ospedali Riuniti di Foggia - U.O.C. di Malattie Infettive, Foggia, Apulia
  - Ospdale San Carlo, Potenza, Basilicate
  - Università della Campania Luigi Vanvitelli - Malattie Infettive, Caserta, Campania
  - A.O.U. Federico II - U.O.C. di Malattie Infettive, Napoli, Campania
  - Azienda Ospedaliera dei Colli - Monaldi Cotugno CTO - IV Divisione, U.O.C. di Immunodeficienze e Malattie Infettive di Genere, Napoli, Campania
  - Presidio Ospedaliero A.O.U. Vanvitelli - U.O. di Malattie Infettive, Napoli, Campania
  - A.O.U. Policlinico S. Orsola-Malpighi, Università degli Studi di Bologna - U.O. di Malattie Infettive, Bologna, Emilia-Romagna
  - BLQ Check Point, Bologna, Emilia-Romagna
  - A.O.U. di Ferrara - Arcispedale Sant'Anna - U.S. Gestione Ambulatorio HIV/AIDS U.O. Malattie Infettive, Ferrara, Emilia-Romagna
  - Università degli Studi di Modena e Reggio Emilia, Modena - Clinica di Malattie Infettive e Tropicali, Modena, Emilia-Romagna
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova - U.O. Malattie Infettive, Reggio Emilia, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Friuli Centrale (ASU FC) Santa Maria della Misericordia - Clinica Malattie Infettive, Udine, Friuli Venezia Giulia
  - Università Sapienza Polo Pontino - U.O. di Malattie Infettive, Latina, Lazio
  - Circolo Mario Mieli, Rome, Lazio
  - INMI "L. Spallanzani" IRCCS - U.O.C. Immunodeficienze Virali, Rome, Lazio
  - Roma Check Point, Rome, Lazio
  - Università Cattolica del Sacro Cuore - Istituto di Clinica delle Malattie Infettive, Rome, Lazio
  - Università degli Studi "La Sapienza" - Dipartimento di Malattie Infettive e Tropicali, Rome, Lazio
  - Università degli Studi di Roma, Policlinico "Tor Vergata" - Divisione di Malattie Infettive, Rome, Lazio
  - Ospedale Bel Colle Viterbo - U.O.C. Medicina protetta - Malattie infettive, Viterbo, Lazio
  - Università di Genova e Ospedale Policlinico San Martino - Clinica di Malattie Infettive, Genoa, Liguria
  - ASST Papa Giovanni XXIII , Struttura Complessa Malattie Infettive, Bergamo, Lombardy
  - Azienda Ospedaliera Spedali Civili di Brescia - I Divisione di Malattie Infettive, Brescia, Lombardy
  - Istituti Ospitalieri di Cremona - U.O. Malattie Infettive, Cremona, Lombardy
  - ASST di Lecco - Ospedale Alessandro Manzoni - S.C. di Malattie Infettive, Lecco, Lombardy
  - Associazione Milano Check Point, Milan, Lombardy
  - ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco - Dipartimento Malattie Infettive, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda - S.C. Malattie Infettive, Milan, Lombardy
  - ASST Santi Paolo e Carlo - U.O.C. di Malattie Infettive e Tropicali, Presidio San Paolo, Milan, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Divisione di Malattie Infettive, Milan, Lombardy
  - Ospedale San Raffaele, Università Vita-Salute - Clinica Malattie Infettive, Milan, Lombardy
  - Ospedale Amedeo di Savoia, Università degli Studi di Torino - Clinica di Malattie Infettive, Turin, Piedmont
  - Policlinico Universitario Duilio Casula, AOU di Cagliari - Medicina Interna e Malattie del Fegato, Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria di Sassari, Malattie Infettive Dipartimento di Medicina Clinica e Sperimentale, Sassari, Sardinia
  - ARNAS Garibaldi - P.O. Nesima - U.O.C. di Malattie Infettive, Catania, Sicily
  - PO "Umberto I" ASP, Enna, Sicily
  - Ospedale Paolo Borsellino - Unità Operativa Complessa Malattie Infettive - ASP, Marsala, Sicily
  - A.O.U. Policlinico "G. Martino" - U.O.C. di Malattie Infettive, Messina, Sicily
  - A.O.U. Policlinico "P. Giaccone" - U.O.C. Malattie Infettive e Centro Regionale di Riferimento AIDS, Palermo, Sicily
  - ARNAS Civico di Cristina Benfratelli - Unità Operativa Malattie infettive, Palermo, Sicily
  - Azienda Sanitaria Provinciale 8 - Presidio Umberto I - U.O. di Malattie Infettive, Syracuse, Sicily
  - A.O.U. Ospedali Riuniti Umberto I - Salesi - Lancisi- Università Politecnica delle Marche Servizio Regionale di Immunologia Clinica e Tipizzazione Tessutale, Ancona, The Marches
  - Azienda Sanitaria dell'Alto Adige - Malattie Infettive, Bolzano, Trentino-Alto Adige
  - Ospedale Santa Chiara di Trento - Unità Operativa di Malattie Infettive, Trento, Trentino-Alto Adige
  - AOUC Azienda Ospedaliero-Universitaria Careggi - S.O.D. di Malattie Infettive e Tropicali, Florence, Tuscany
  - Ospedale Santa Maria Annunziata - Azienda Sanitaria di Firenze - U.O. di Malattie Infettive, Florence, Tuscany
  - Presidio Ospedaliero di Pistoia - U.O. Malattie Infettive II, Pistoia, Tuscany
  - A.O.U. Senese, Policlinico S. Maria alle Scotte - U.O.C. di Malattie Infettive, Siena, Tuscany
  - Azienda Ospedaliera di Padova - U.O.C. Malattie Infettive, Padua, Veneto
  - Azienda ULSS 8 Berica - Divisione Malattie Infettive, Vicenza, Veneto

IPD SHARING:
Plan to Share IPD: No